CLINICAL TRIAL: NCT05080855
Title: Unilateral Cleft Lip Repair: Quantitative (Anthropometric) Comparative Assessment of Modified Millard vs Tennison-Randall Techniques.
Brief Title: Comparison of Techniques in Repair of Unilateral Cleft Lip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Salah Ahmed, Faculty of Pediatric Surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150318
Record Dates: First submitted 2021-09-28; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Unilateral Cleft Lip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the cleft lip will be repaired by modified Millard technique (Active Comparator): In the modified Millard technique, points (nasal and Vermilion border points) and lines (rotational and advancement flap lines and mucosal lines) were drawn. Then, we cut the submucosal layer and created three flaps: advancement flap, rotational flap, and c flap. The orbicular muscle was dissected and freed from the columellar base on the non-cleft side and from the alar base on the cleft side. Using a vicryl 5-0, we sutured the anterior nasal floor; then, using vicryl 4-0, we sutured the alar base and muscle. Using vicryl 6-0, we sutured top of philtral column with point a, the peak of Cupid's bow, and tip of c flap with alar base. The suturing of mucosal lip was carried out using a vicryl 5-0.
  Interventions: Procedure: modified Millard technique vs Tennison-Randall technique
- the cleft lip will be repaired by Tennison-Randall technique. (Active Comparator): In the Tennison-Randall technique, points (nasal and Vermilion border points) and lines (Skin triangle flap lines and mucosal lines) were drawn. Then, we cut the submucosal layer and created equilateral triangle flap and releasing incision. The orbicular muscle was dissected and freed from the columellar base on the non-cleft side and from the alar base on the cleft side. The suturing of the anterior nasal floor, alar base, and muscle followed the same principles of the modified Millard technique. The cutaneous repair was done by suturing the top of philtral column, the peak of Cupid's bow, point a, the line between the top of philtral column and the peak of Cupid's bow with b-8 and 3-a with b-a.
  Interventions: Procedure: modified Millard technique vs Tennison-Randall technique

INTERVENTIONS:
Procedure: modified Millard technique vs Tennison-Randall technique — evaluate the quantitative (anthropometric) assessment of modified Millard technique in comparison to Tennison-Randall technique in unilateral cleft lip (ucl) repair. Inclusion criteria: Patient with ages from 2 months old to 6 months old, Patient with unilateral cleft lip complete or incomplete type.

SUMMARY:
Over the past century, there have been major advances in unilateral cleft-lip repair techniques toward the method's modern form. The first documented cleft-lip repair involved simple freshening and approximation of the cut cleft edges, followed by the use of curved incisions to allow lengthening of the lip. Straight-line closure repairs were used in the early 1900; however, straight-line closures had the disadvantage of creating a vertical scar contracture, leading to notching of the lip. This led to the development of several methods in the mid-twentieth century that are grouped as quadrangular flaps, triangular flaps, and rotation-advancement techniques.

The two basic techniques that are most commonly used for unilateral cleft lip (UCL) closure are the Tennison-Randall and the Millard rotation_advancement techniques. both techniques address the importance of repositioning the lip muscle (orbicularis oris) in the correct anatomic orientation for optimal aesthetic and functional outcomes.

The ultimate goal of cleft lip surgery is to achieve a perfectly symmetrical lip and nose. It has been shown that for the general population, the more symmetrical the face, the more attractive the face is. The appearance and symmetry of the nasolabial region is also seen as one of the most important characteristics when evaluating the results of any facial surgery.

Measurement of treatment outcome is vital to evaluate the success of cleft management and the degree of improvement, especially in the present age of evidence-based medicine where treatment guidelines for best practice are becoming an integral part of contemporary clinical practice.

The good goal of cleft lip repair is a symmetrical and balanced lip with minimal scar restoring the natural contours of the face, as well as correcting functional anatomy.

Objectives To evaluate the quantitative (anthropometric) assessment of modified Millard technique in comparison to Tennison_ Randall technique in unilateral cleft lip (ucl) repair.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with age from 2 months old to 6 months old.
2. Patient with unilateral cleft lip complete or incomplete type.

Exclusion Criteria:

1. Patient with age less than 2 months old or more than 6 months old.
2. Patients with bilateral cleft lip
3. Patients with recurrent cleft lip.
4. Patients with associated major congenital anomalies like major cardiac anomalies.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Assessment of Post-operative Complications | 1 month
  Early:
  Wound infection. Wound dehiscence.
  Late:
  Wound scarring. Lip notch

SECONDARY OUTCOMES:
Anthropometry assessment of Cosmetic Results | patients were assessed before the operation and followed for 3-4 weeks after.
  Anthropometric measurements were recorded from a two dimensional full-frontal facial photograph of subjects will be taken with a digital camera. The following anthropometric measurements will be taken. Preoperative(measurements will be taken before the surgery).
  Vertical lip height on( both cleft and non-cleft side), Horizontal lip length on( both cleft and non-cleft side), Nasal width, Total nasal width.
  Postoperative (measurements will be taken three months after the surgery). Vertical lip height on( both cleft and non-cleft side), Horizontal lip length on( both cleft and non-cleft side), Nasal width, Total nasal width.
Satisfaction score | 24 hours after the operation
  by patient parent's satisfaction.
Operative time | intraoperatively
  from the first landmark design to the last suture.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Surgery department, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No